CLINICAL TRIAL: NCT06106620
Title: Effects of a Multi-Ingredient Dietary Supplement Consisting of Vitamins, Minerals, Botanicals, and Nootropics on Blood and Breath Alcohol Levels
Brief Title: Effects of a Multi-Ingredient Dietary Supplement on Blood and Breath Alcohol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SS-1023-001
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 12 oz of flavor-matched water.
  Interventions: Dietary Supplement: Placebo
- Safety Shot (Experimental): 12 oz of Safety Shot containing a blend of vitamins, minerals and botanical extracts.
  Interventions: Dietary Supplement: Safety Shot

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo drink consisting of 12 oz of flavor-matched water.
  Arms: Placebo
Dietary Supplement: Safety Shot — Safety Shot consisting of a 12 oz drink containing vitamins, mineral, and botanical extracts.
  Arms: Safety Shot

SUMMARY:
This study is a randomized, two-arm, double-blind, placebo-controlled, crossover study of N=36 apparently healthy men and women. This study will assess the effect of a blend of dietary supplements on blood and breath levels after consuming alcohol.

DETAILED DESCRIPTION:
This study is a randomized, two-arm, double-blind, placebo-controlled, crossover study of N=36 apparently healthy men and women. This study will assess the effect of a blend of dietary supplements on blood and breath levels after consuming alcohol. Consumption of this dietary supplement is not intended to diagnose, treat, cure, or prevent any disease.

Participants will attend three study visits. During Visit 1, participants will be screened for participation (i.e., medical history, routine blood work, and background baseline diet. During Visits 2 and 3 participants will ingest 100 mL (3.4 oz) of 40% alcohol, along with a commercially available liquid blend of dietary supplements or a placebo, and undergo assessments of breath alcohol content, blood alcohol levels, blood alcohol dehydrogenase levels, and various visual analog scales (VAS) for indices of affect (headache, nausea, fatigue, energy, tiredness, thirst, concentration) for 4 hours post-ingestion. Safety will be monitored via vital signs (heart rate, blood pressure) and adverse events (AE) throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 21 and 55 (inclusive).
* Body Mass Index of 18.5-34.9 (inclusive).
* Body weight of at least 110 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from alcohol for 48 hours, caffeine and exercise for 24 hours prior to each trial, and fast for 10 hours prior each of the treatments.
* Agreeable to have a third-party transport home following interventional visits.
* Able to provide an adequate blood draw.
* Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
* Subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal disease.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or history of drug/alcohol abuse or dependence.
* History of diabetes or endocrine disorder.
* Fasting blood sugar of > 125 mg/dL.
* Current smokers or cessation of smoking within the past month.
* History of hyperparathyroidism or an untreated thyroid disease.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc., known gastrointestinal disorder that may impact nutrient absorption e.g., short bowel syndrome, atrophic gastritis, IBD, diarrheal illnesses, history of colon resection, gastro-paresis, celiac disease, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g., rheumatoid arthritis, Crohn's Disease, ulcerative colitis, lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women. Women who participate in this study must agree to the use of contraception for the duration of the study and any woman that is sexually active will have to take a negative pregnancy test prior to enrolling. Women of childbearing age (any woman prior to menopause) regardless of their use of contraception will be provided a urine pregnancy test kit at their screening visit and take the test in private using the female lavatory after signing an informed consent.
* Known sensitivity to any ingredient in the test formulations as listed in the product label.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Headache | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Headache as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent a greater headache.
Nausea | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Nausea as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater nausea.
Fatigue | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Fatigue as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater fatigue.
Energy | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Energy as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater energy.
Tiredness | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Tiredness as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater tiredness.
Thirst | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Thirst as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater thirst.
Concentration | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Concentration as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater concentration.

SECONDARY OUTCOMES:
Breath alcohol level | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Breath alcohol level measured in %.
Blood alcohol level | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Blood alcohol level measured in milligrams per deciliter (mg/dL).
Blood alcohol dehydrogenase level | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Blood alcohol dehydrogenase level measured picograms per milliliter (pg/mL).
Blood acetaldehyde level | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Blood acetaldehyde level as measured in milligrams per deciliter (mg/dL).
Blood aldehyde dehydrogenase level | Change from baseline to 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Blood aldehyde dehydrogenase level as measured in nanograms per milliliter (ng/mL).
Urine volume | Change from baseline to 60 minutes, 120 minutes, 180 minutes, and 240 minutes.
  Urine volume as measured in milliliters.

OTHER OUTCOMES:
Systolic blood pressure | Change from baseline to 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Systolic blood pressure in mm of mercury.
Diastolic blood pressure | Change from baseline to 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Diastolic blood pressure in mm of mercury.
Heart rate | Change from baseline to 60 minutes, 120 minutes, 180 minutes and 240 minutes.
  Heart rate in beats per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided